CLINICAL TRIAL: NCT04617405
Title: Hormonal and Inflammatory Changes During Pregnancy in Women With Glucose Metabolic Disorders.
Acronym: HI-MET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: PADME1
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2; Gestational Diabetes; Overweight and Obesity; Pregnancy in Diabetic; Insulin Resistance; Insulin Sensitivity; Pregnancy, High Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Overweight; Obesity; Pregnancy in Diabetics; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type A: Healthy normal-weight pregnant women
  Interventions: Other: No interventions
- Type B: Pregnant women with gestational diabetes diagnosed at early screening (before gestational week 20)
  Interventions: Other: No interventions
- Type C: Pregnant women with type 2 diabetes
  Interventions: Other: No interventions
- Type D: Healthy overweight pregnant women
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
The first aim of this study is to describe maternal hormonal and inflammatory changes during pregnancy in women that differ metabolically (limited to women with type 2 diabetes, gestational diabetes and/or overweight). The second aim of this study is to examine maternal hormonal, inflammatory and metabolic factors associated with insulin sensitivity in human pregnancy.

DETAILED DESCRIPTION:
This is a prospective observational study including app. 300 pregnant women from the outpatient clinics at Department of Obstetrics and Gynecology at Aalborg, Odense and Aarhus University Hospital.

The study includes 50 healthy normal-weight women, 150 healthy overweight women, 50 women with gestational diabetes and 50 women with type 2 diabetes.

Hormonal profiles and inflammatory markers will be measured at gestational week 8-10, 10-14, 18-22, 24-28 and 34-38. The blood samples will include HbA1c, glukose, insulin, C-peptid, lipid profile, liver enzymes, creatinine, FGF-21, TSH, Cortisol, human chorionic gonadotropin, estradiol, progesterone, prolactin, human placental lactogen, placental growth hormone, IGF-1, IGF-BP's, Leptin, Adiponectin, GLP-1, GIP, hs-CRP, IL-6, IL-10, IL-1α, IFN-ɣ, TNF-α, ICAM1, VCAM and CD163. In addition to this, exosomes will be isolated precisely and profiling of the content of exosomes will be performed using in vitro assays. Proteomics and miRNAs sequencing will be employed.

Height, weight, and blood pressure will be measured at every visit and a urine sample will be collected.

Insulin sensitivity will be estimated using the homeostasis model assessment, IS-HOMA, based on fasting insulin and glucose concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at The Department of Gynaecology and Obstetrics at Aarhus University Hospital, Aalborg University Hospital or Odense University Hospital.
* Women have to be in 1 of 4 categories: Healthy with a BMI < 25, healthy with a BMI >= 25, diagnosed with gestational diabetes before gestational week 20 or diagnosed with pregestational type 2 diabetes

Exclusion Criteria:

* Age < 18 years
* Not able to read and understand danish
* Previous bariatric surgery
* Treatment with systemic corticosteroids

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are eligible for participation.
Study Population: The study population consist of pregnant women followed at The Department of Gynaecology and Obstetrics at Aarhus University Hospital, Aalborg University Hospital or Odense University Hospital. Cases are either healthy with a BMI >= 25, diagnosed with gestational diabetes before gestational week 20 or diagnosed with pregestational type 2 diabetes. Controls are healthy with a BMI < 25.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in serum or plasma concentration of metabolic, hormonal and inflammatory markers at four other times during pregnancy. | Gestational week 8-10 (baseline), gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Serum concentration of IGF-1, IGFBP-3, IGFBP-1, FGF-21, Leptin, Adiponectin, CD163, Human Chorionic Gonadotropin, Progesterone, C-peptide, Cortisol, Prolactin, Sex Hormone Binding Globulin, Estradiol, Free fatty acids, Human Placental Lactogen and Human Placental Growth Hormone.
  Plasma concentrations of IL-6, IL-10, IL-1alpha, IFN-gamma, TNF-alpha, ICAM1, VCAM, LDL, HDL, Triglyceride, Gamma-Glutamyl Transferase, Thyrotropin, glucose and HbA1c.
Assocation between the serum or plasma concentration of metabolic, hormonal and inflammatory markers Versus Insulin sensitivity at five times during pregnancy. | Gestational week 8-10, gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Association between the metabolic, hormonal and inflammatory markers listed as Primary Outcome 1 and the Insulin sensitivity. Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting insulin and glucose concentrations.
Changes from baseline in the level, content and bioactivity of exosomes in serum and plasma at four other times during pregnancy. | Gestational week 8-10 (baseline), gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Exosomes will be isolated and profiling of the content will be performed using SWATH mass spectrometry and miRNA sequencing.
Association between the level, content and bioactivity of exosomes in serum and plasma Versus Insulin sensitivity at five times during pregnancy. | Gestational week 8-10, gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Exosomes will be isolated and profiling of the content will be performed using SWATH mass spectrometry and miRNA sequencing. Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting insulin and glucose concentrations.

SECONDARY OUTCOMES:
Changes from baseline in blood pressure (systolic and diastolic) at four other times during pregnancy. | Gestational week 8-10 (baseline), gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Blood pressure includes the measurement of both systolic and diastolic blood pressure (mmHg).
Changes from baseline in body weight at four other times during pregnancy. | Gestational week 8-10 (baseline), gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Body weight measured in kilograms.
Association between the blood pressure (systolic and diastolic) Versus Insulin sensitivity at five times during pregnancy. | Gestational week 8-10, gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Blood pressure includes the measurement of both systolic and diastolic blood pressure (mmHg). Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting insulin and glucose concentrations.
Association between the body weight Versus Insulin sensitivity at five times during pregnancy. | Gestational week 8-10, gestational week 10-14, gestational week 18-22, gestational week 24-28 and gestational week 34-38
  Body weight measured in kilograms. Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting insulin and glucose concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Koefoed, M.D., Principal Investigator — Aarhus University, Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No